CLINICAL TRIAL: NCT00176319
Title: Age-related Functional and Molecular Effects of Short-term Aerobic Endurance Training in Patients With Stable Chronic Heart Failure and Age-matched Healthy Controls.
Brief Title: Leipzig Exercise Intervention in Chronic Heart Failure and Aging
Acronym: LEICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GI 535/1-1; GI 535/1-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Heart Failure; Ageing
Keywords: heart failure; ageing
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Behavioral: Aerobic endurance exercise training (ergometer)

SUMMARY:
In both ageing and heart failure progressive exercise intolerance is observed. The Leipzig Exercise Intervention in Chronic heart failure and Aging (LEICA) study aims to investigate how aerobic short-term training interventions affect exercise capacity, left ventricular systolic and diastolic function, biomarkers of heart failure, skeletal muscle metabolism, and endothelial function in chronis heart failure patients (CHF-patients) and healthy subjects (HS) in two different age strata: Above 65 years and below 55 years.

Aim of the trial is therefore to compare the effects of aerobic exercise training in young and old healthy subjects as well as in young and old heart failure patients. To our knowledge this study is the first to prospectively investigate age differences of training responses in both CHF patients and age-matched healthy controls.

Because of the extensive clinical and molecular assessment the results of this trial will be made public in predefined substudies:

* LEICA-Echo
* LEICA-Biomarkers
* LEICA-Endothelium
* LEICA-Cardiopulmonary Exercise Function
* LEICA-Muscle

DETAILED DESCRIPTION:
A total of 60 healthy subjects and 60 heart failure patients (in each group 30 <55 years, 30 >65 years) are prospectively randomized to either 4 weeks of aerobic ergometer training or control group.

Before and after the intervention period maximal exercise tolerance is determined by ergospirometry, endothelial function is measured by high-resolution A-mode ultrasound, left ventricular function by echocardiography including tissue Doppler imaging, and thigh muscle mass is assessed by CT. Skeletal muscle biopsies are obtained at both time-points and are analysed for inflammatory cytokines and markers of catabolism/anabolism.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Healthy subjects

* normal left ventricular ejection fraction (EF) >55%
* normal coronary artery disease (cardiac catheterization)

Group 2: CHF patients

* reduced left ventricular ejection fraction (EF) <40%
* stable clinical condition (NYHA II-III)

Exclusion Criteria:

* COLD
* cardiac decompensation <3 months
* ventricular arrhythmias >Lown IVb
* myocardial infarction < 4 weeks
* valvular heart disease >II°
* insulin-dependent diabetes mellitus
* arterial hypertension
* orthopedic conditions prohibiting training participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Improvement in functional exercise capacity (as measured by cardiopulmonary exercise testing)
Echocardiography: Improvement in left ventricular diastolic function as assessed by tissue Doppler (E/E' ratio)

SECONDARY OUTCOMES:
Biomarkers of heart failure (including NT-proBNP)
Endothelial function
Activation of the catabolic ubiquitin-proteasome pathway

CONTACTS AND LOCATIONS:
Overall Officials: Rainer P Hambrecht, MD, Principal Investigator — University of Leipzig, Heart Center, Dept. of Cardiology; Stephan Gielen, MD, Principal Investigator — University of Leipzig - Heart Center, Dept. of Internal Medicine/Cardiology; Volker Adams, PhD, Study Director — University of Leipzig, Heart Center, Dept. of Internal Medicine/Cardiology
Locations (1):
- Universität Leipzig, Herzzentrum, Klinik für Innere Medizin/Kardiologie, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Gielen S, Sandri M, Kozarez I, Kratzsch J, Teupser D, Thiery J, Erbs S, Mangner N, Lenk K, Hambrecht R, Schuler G, Adams V. Exercise training attenuates MuRF-1 expression in the skeletal muscle of patients with chronic heart failure independent of age: the randomized Leipzig Exercise Intervention in Chronic Heart Failure and Aging catabolism study. Circulation. 2012 Jun 5;125(22):2716-27. doi: 10.1161/CIRCULATIONAHA.111.047381. Epub 2012 May 7. PMID 22565934
- [Derived] Sandri M, Kozarez I, Adams V, Mangner N, Hollriegel R, Erbs S, Linke A, Mobius-Winkler S, Thiery J, Kratzsch J, Teupser D, Mende M, Hambrecht R, Schuler G, Gielen S. Age-related effects of exercise training on diastolic function in heart failure with reduced ejection fraction: the Leipzig Exercise Intervention in Chronic Heart Failure and Aging (LEICA) Diastolic Dysfunction Study. Eur Heart J. 2012 Jul;33(14):1758-68. doi: 10.1093/eurheartj/ehr469. Epub 2012 Jan 19. PMID 22267243